CLINICAL TRIAL: NCT06953609
Title: Effects of Prediabetes and Type 2 Diabetes on Cognitive Status, Physical Function, and Fatigue in Geriatric Individuals: A Case-Control Study
Brief Title: Prediabetes and Type 2 Diabetes in Aging
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Kevser Gürsan, Principal Investigator, Uşak University
Other Study IDs: 562-562-11
Record Dates: First submitted 2025-04-19; First posted 2025-05-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Cognitive Function; Dual Task; Fatigue; Prediabetes
Keywords: type 2 diabetes mellitus; cognitive function; dual task; fatigue; prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatigue; Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: The normal range for Hemoglobin A1c Levels (HbA1c) for people without diabetes (Healthy) is those with an HbA1c level between 4% and 5.6%,
- A prediabetes (Impaired Glucose Tolerance): those with a prediabetes (Impaired Glucose Tolerance) level between 5.7% and 6.4%
- Those with type 2 DM (controlled): those with a HbA1c Levels of 6.5% - 7.5%
- Those with type 2 DM (uncontrolled): those with an HbA1c level above 7.5

SUMMARY:
This case-control study will evaluate the effects of geriatric individuals on cognitive status, physical function and fatigue. Our study aims to compare the effects of geriatric individuals with prediabetes and type 2 diabetes with healthy geriatric individuals on cognitive status, physical function and fatigue. Accordingly, the hypotheses of the study are as follows:

Hypothesis 1: Prediabetes and Type 2 Diabetes Negatively Affect Cognitive Status in Geriatric Individuals.

Hypothesis 2: Physical Function Loss is More Pronounced in Individuals with Prediabetes and Type 2 Diabetes.

Hypothesis 3: Fatigue Level Will Increase in Geriatric Individuals with Prediabetes and Type 2 Diabetes.

Hypothesis 4: There Will Be a Correlation Between the Effects of Prediabetes and Type 2 Diabetes on Cognitive Status, Physical Function and Fatigue.

Hypothesis 5: Severity of Diabetes (Prediabetes vs. Type 2 Diabetes) Will Create Differences in Cognitive, Physical and Fatigue Status.

Prediabetic, diabetic and healthy volunteers constitute the universe of the study. There will be 4 different groups in the study. These groups are; those with normal range of Hemoglobin A1c Levels (HbA1c) between 4% and 5.6% for people without diabetes (Healthy), those with HbA1c level between 5.7% and 6.4%, those with prediabetes (Impaired Glucose Tolerance), those with 6.5% - 7.5% and those with HbA1c level above 7.5. Cognitive status, physical functions, dual task performance, motor motor and motor cognitive performances, fatigue, reaction reactions, directional skills of elderly individuals will be compared between these groups.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus develops due to insulin resistance and/or decreased insulin secretion and is particularly common in the elderly population. With the aging process, metabolic changes and increased insulin resistance increase the risk of diabetes. Long-term complications of diabetes can negatively affect the quality of life in geriatric individuals with effects such as cognitive impairment, loss of physical function and fatigue. In individuals with diabetes, hyperglycemia, microvascular complications and inflammation can increase the risk of cognitive decline. This can pave the way for dementia and Alzheimer's disease. Prediabetes is a condition in which blood sugar levels are higher than normal, but not high enough to diagnose diabetes, and this is an important risk factor for Type 2 Diabetes Mellitus. Even prediabetes has been associated with deterioration in cognitive functions. Loss of muscle mass (sarcopenia) and decreased physical endurance are frequently seen in geriatric individuals with diabetes. These individuals are likely to experience mobility problems and have an increased risk of falling. Chronic fatigue is another common complication of diabetes. Hyperglycemia can affect energy metabolism and cause fatigue. Fatigue can reduce physical activity levels and worsen general health status. Based on this, the study will include 4 groups: geriatric individuals with prediabetes and type 2 diabetes (controlled and uncontrolled) and healthy geriatric individuals. It will be compared whether there are any differences between these groups in terms of cognitive status, reaction times, sense of direction, dual task performance, physical function and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* for people without diabetes (healthy), those with Hemoglobin A1c Levels (HbA1c) normal range between 4% and 5.6%,
* those with HbA1c level between 5.7% and 6.4%, those with prediabetes (Impaired Glucose Tolerance),
* those with 6.5% -7.5% level and
* those with HbA1c level above 7.5
* criteria are being 60 years of age and older,

Exclusion Criteria:

* those who have major depression,
* uncontrolled thyroid disease,
* those with vitamin B12, folic acid deficiency and anemia,
* those with uncontrolled hypertension,
* those with nephropathy and retrophy,
* those with any neuropsychological disorder, a history of alcohol, substance or drug addiction,
* those using any neurological or psychological medication (anticonvulsant drugs, antidepressants, anxiolytics, etc.),
* those with Alzheimer's and Parkinson's disease,
* those with cancer,
* those with lung disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in 4 different Endocrinology clinics in Uşak, Turkey. Approximately 80 patients and healthy volunteers who meet the inclusion criteria for the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Cognitive status assessment | At the time of enrollment
  The cognitive status of elderly individuals will be assessed with the Montreal Cognitive Assessment test. MoCA is a neuropsychological test developed to assess mild cognitive impairment (MCI) and early-stage dementia. It is evaluated out of 30 points and a score of 26 and above is considered normal. Validity and reliability in Turkish have been performed.

SECONDARY OUTCOMES:
Assessing sense of direction. | At the time of enrollment
  Santa Barbara Sense of Direction Scale (SBSOD): It is a self-report scale that assesses the ability of individuals to find their way. It assesses components such as wayfinding competence, internal mapping skills, and environmental cognition. Scale structure: It usually consists of 15 items and is assessed with a Likert-type score between 1-7. Subtests: It includes visual-spatial skills, short-term memory, attention, concentration, working memory, language, and orientation.
Reaction evaluation | At the time of enrollment
  The Nelson Foot Reaction Test will be used to evaluate the reaction. Nelson Foot Reaction Test: It is a test that measures the reaction time to visual stimuli. In the foot reaction test, the ruler is placed between the fingers.
  The operator holds the ruler from its tip and up. After giving the ready signal, he/she releases the ruler for a while. The subject tries to catch the ruler as soon as possible. The reaction time is calculated according to the distance at the point he/she caught and recorded.
Assessment of Blood glucose | At the time of the enrollment
  Blood glucose (mg/dL) - To explore the relationship between glycemic status and fatigue.
Assessment of Cortisol (µg/dL) | At the enrollment
  Cortisol (µg/dL) - Morning cortisol levels will be assessed as an indicator of adrenal function and fatigue.
Dual task performance assessment | At the time of enrollment
  To assess dual task performance, both motor-motor and motor-cognitive tasks will be assessed.
  Cognitive-Motor Task: Walking 3 meters while counting the days of the week backwards, assesses the interaction between walking and cognitive workload.
  Motor-Motor Task: Walking 3 meters while carrying 4 water bottles, assesses postural control and motor coordination
Physical Function Assessment | At the time of enrollment
  A distance of 3 meters is measured for the starting and returning points and this distance is taped. The patient is seated in a chair next to the starting line The procedure is explained to the patient The patient is asked to walk to the mark 3 meters away, turn around and sit back in the chair. The elapsed time is recorded with a stopwatch.
Self-report assessment of fatigue | At the time of enrollment
  Fatigue is measured with both subjective scales. Self-report assessment of fatigue will be made with the fatigue severity scale.Fatigue Severity Scale is used to assess the level of fatigue of individuals in their daily life activities. It consists of 9 items and is scored between 1-7.
Assessment of Hemoglobin level | At the time of enrollment
  Hemoglobin level (g/dL) - Blood samples will be collected to measure the participants' hemoglobin concentration to evaluate fatigue-related anemia.
Assessment of Serum ferritin | At the time of enrollment
  Serum ferritin (ng/mL) - To assess iron stores which may influence fatigue levels.
Assessment of Thyroid stimulating hormone (TSH) | At the time of enrollment
  Thyroid stimulating hormone (TSH) (µIU/mL) - To evaluate thyroid-related causes of fatigue.
Assessment of C-reactive protein (CRP) | At the time of enrollment
  C-reactive protein (CRP) (mg/L) - As a marker of systemic inflammation related to fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Gursan, Dr., Principal Investigator — Uşak University
Locations (1):
- Uşak Education and Research Hospital, Uşak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect participant confidentiality and comply with the confidentiality commitment approved by the ethics committee, no sharing of individual-level data is planned. In addition, the ethics committee decision that approved the study covers data use with limited access only. Therefore, it may not be possible to share IPD data publicly.